CLINICAL TRIAL: NCT04587739
Title: A Pilot Study on the Feasibility and Tolerance of Neoadjuvant Hypofractionated, Stereotactic Body Radiation Therapy Prior to Surgical Resection of Uninodular Hepatocellular Carcinoma.
Brief Title: Neoadjuvant Hypofractionated Stereotactic Body Radiation Therapy Prior to Surgery for Hepatocellular Carcinoma: a Feasibility Study.
Acronym: KARCHER-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017_03; 2019-A01441-56 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-10-13; First posted 2020-10-14 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Stereotactic body radiation therapy; Hepatectomy; Neoadjuvant therapy; Drop-out
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Combination Product: Surgery with Neoadjuvant stereotactic body radiation therapy

INTERVENTIONS:
Combination Product: Surgery with Neoadjuvant stereotactic body radiation therapy — Stereotactic hypofractionated robotic radiation therapy (24-45 Gy / 3 fractions) followed after 4-6 weeks by conventional hepatectomy (either anatomical liver resection, or non-anatomical liver resection with intention to achieve a minimal 2 cm margin).

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth more common cancer in the world, with high mortality rates, due to the low number of patients who are eligible for therapy with curative intent, like surgical resection. Moreover, surgical resection is associated with a high risk of tumor recurrence, because of the tumor seeding through microscopic intrahepatic vessels that surround the tumor, the so-called "microvascular invasion".

To adequately deal with this phenomenon, the surgeon has to perform either an 'anatomical' liver resection, which remove not only the tumor but also the whole corresponding vascular network, or a 'tumorectomy' with resection margins of at least 2 cm. Unfortunately, these principles cannot always be achieved due to underlying liver cirrhosis that is present in more than 80% of patients.

Stereotactic body radiation therapy (SBRT) has been proven to efficiently necrotize or stabilize HCC nodules when surgery is not possible. Our hypothesis is that pre-treatment with SBRT prior to surgical resection of HCC might improve the results through the destruction of possible seeding in the peritumoral environment.

Given the novelty of this therapeutic strategy, it is necessary to verify its feasibility and safety, prior to test its efficacy in patients with HCC. The KARCHeR-1 study aims at making sure that preoperative SBRT would not result in important delays or serious adverse events such as to cancel the planned surgical resection, in patients who otherwise could have benefited from it. This issue is commonly called 'drop-out'. Thirty patients are expected to be included in the KARCHeR-1 study, which would be in favor of continuing to evaluate this therapeutic strategy if less than 3 drop-outs occur, and would be immediately discontinued if 3 drop-outs occur. Other outcomes will also been studied, like intraoperative issues, postoperative morbi-mortality, pathological features on the surgical specimen and its correlation with preoperative imaging, and finally, tumor recurrence and survival.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven hepatocellular carcinoma or EASL/AASLD criteria
* Single nodule, 3 to 8 cm of largest diameter
* Hepatocellular carcinoma eligible for conventional liver resection with curative intent (R0), without preoperative portal vein embolization

Exclusion Criteria:

* Performance status > 2
* Severe comorbidity with contraindication for either surgery or radiation therapy
* Decompensated liver cirrhosis (Child-Pugh B or C)
* Neoplastic portal vein thrombosis or extra-hepatic metastases
* Previous anticancer therapy within the last 5 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-31 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Drop-out rate | Five months after the inclusion of the last participating patient
  Drop-out rate: proportion of patients in whom surgical resection cannot be achieved, due to (at least one of the following reasons):
  * serious adverse events related to radiation therapy (especially liver decompensation);
  * disease progression while receiving radiation therapy or awaiting surgery;
  * patient's death.

SECONDARY OUTCOMES:
Intraoperative number of packed red blood cells transfused (if any). | Postoperative 90 days
Toxicity of radiation therapy using the National Cancer Institute CTCAE v.5.0 criteria | Postoperative 90 days
Duration of surgery. | Postoperative 90 days
Volume of intraoperative blood loss | Postoperative 90 days
Quality of life by EORTC QLQ-C30 | between before and after stereotactic radiotherapy
Intraoperative adverse events | Postoperative 90 days
Postoperative severe and overall morbidity rate | Postoperative 90 days
  defined using the Comprehensive Complication Index and graded with the Dindo-Clavien score
Postoperative mortality rate. | Postoperative 90 days
Correlation between radiological observations on preoperative imaging and pathological features on surgical specimen (like percentage of tumor necrosis). | Postoperative day 30.
Actuarial overall survival and disease-free survival. | Postoperative 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Boleslawski, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France